CLINICAL TRIAL: NCT02883816
Title: Early Assessment of Respiratory Function, Inflammation and Bronchial Reshuffle Among Newborns Screened for Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8229
Record Dates: First submitted 2016-08-09; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cystic fibrosis (Experimental): assessment of lung function in newborns screened for cystic fibrosis
  Interventions: Other: assessment of lung function

INTERVENTIONS:
Other: assessment of lung function — measurement of lung volumes and flow rates of bronchial

SUMMARY:
The main objective of this study is to show that there is a concordance between lung disease at 13 months and the existing 9 weeks in newborn babies with cystic fibrosis asymptomatically.

This will identify at the first examination at 8 weeks, newborns who have the most impaired lung function at 13 months. To meet this objective an assessment of their lung function at 9 weeks and 1 month will be performed in newborns diagnosed with cystic fibrosis.

ELIGIBILITY:
Inclusion criteria :

* Infant aged 11 weeks

Exclusion criteria :

* Gestational age lower than 35 weeks of gestation,
* Background invasive mechanical ventilation in positive pressure
* Documented -Obstructive Sleep Apnea, heart defect, neuromuscular disease

Ages: 8 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2008-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from respiratory function at 7 months and 11 months | 7 months and 11 months
  measurement of lung volumes and flow rates of bronchial

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France